CLINICAL TRIAL: NCT07275593
Title: Comparison of Outcome Between Dexamethasone Versus Prednisolone Administration in Acute Exacerbation of Childhood Asthma
Brief Title: Dexamethasone Versus Prednisolone in Acute Exacerbation of Childhood Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR-ASIF-MULTAN
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Exacerbation of Asthma
MeSH Terms: interventions — Dexamethasone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Dexamethasone Group (Experimental): Patients received a single IV dose of dexamethasone at a dose of 0.6 mg/kg.
  Interventions: Drug: Dexamethasone
- Oral Prednisone Group (Experimental): Patients were given oral prednisone at a dose of 2 mg/kg/day (max 60 mg) as a single dose for 3 days.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Dexamethasone — Patients received single IV dose of Dexamethasone at a dose of 0.6 mg/kg
  Arms: Intravenous Dexamethasone Group
Drug: Prednisolone — Patients received oral prednisone at a dose of 2 mg/kg/day (max 60 mg) as a single dose for 3 days.
  Arms: Oral Prednisone Group

SUMMARY:
Because of insufficient local comparative data, this study was designed to determine the outcome of intravenous dexamethasone in contrast to oral prednisolone in acute exacerbation of asthmatic children.

DETAILED DESCRIPTION:
The findings of this study would furnish the local data. The results would also provide recommendations to use more appropriate steroid options in the local settings, resulting in aid to improve the quality of life of asthmatic children and their quicker return to daily routine activities.

ELIGIBILITY:
Inclusion Criteria:

* Children of any gender
* Aged 2-12 years
* Presenting with acute exacerbation of asthma within 24-hours

Exclusion Criteria:

* Children with PRAM score of ≥ 10
* Used oral or parenteral corticosteroids in last 4-weeks
* With any chronic condition of lungs (TB, cystic fibrosis), liver (chronic liver disease), kidneys (chronic kidney disease, nephrotic syndrome) or blood (thalassemia, malignancy)

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2024-11-03 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbation | 4 days
  The Pediatric Respiratory Assessment Measure (PRAM) score was used to assess the severity of asthma exacerbation. This score consisted of 5 items and had a maximum score of 12: suprasternal retractions (0-2), scalene muscle contraction (0-2), air entry in chest (0-3), wheeze (0-3), and oxygen saturation (0-2). A score of 1-3 showed mild exacerbation, 4-7 showed moderate exacerbation, and 8-12 revealed severe exacerbation of asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Asif Abrar, Principal Investigator — Nishter Hospital Multan, Pakistan; Azam Khan, Study Director — Nishter Hospital Multan, Pakistan
Locations (1):
- Nishtar Medical University Hospital, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.